CLINICAL TRIAL: NCT00095784
Title: A Phase II Study of Decitabine in Myelofibrosis
Brief Title: Decitabine in Treating Patients With Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01444; NCI-2011-01444 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000393839; NCI-6814; UCCRC-13327A; 13327A (Other: University of Chicago Comprehensive Cancer Center); 6814 (Other: CTEP); N01CM62201 (NIH); N01CM62207 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Decitabine; Injections

ARMS (1):
- Treatment (decitabine) (Experimental): Patients receive decitabine SC on days 1-5 and 8-12. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Decitabine — Given SC
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well decitabine works in treating patients with myelofibrosis, a cancer of the blood system associated with fibrosis (scar tissue) in the bone marrow that is advanced and for which there is no standard therapy. Decitabine may block the actions of some proteins that are responsible for turning certain genes off in various cancers including myelofibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine response rate (complete and partial responses and hematological improvement) to decitabine in patients with myelofibrosis.

II. To determine the safety of decitabine in patients with myelofibrosis.

SECONDARY OBJECTIVES:

I. To determine the effects of decitabine on specific epigenetic changes including methylation status of specific target genes and gene re-expression.

II. To determine the effect of decitabine on hemoglobin F levels and on the absolute numbers of circulating cluster of differentiation (CD) 34+ progenitor cells and to investigate the potential utility of these markers as a surrogate for biologic activity of decitabine in myeloid metaplasia with myelofibrosis (MMM).

OUTLINE:

Patients receive decitabine subcutaneously (SC) on days 1-5 and 8-12. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed myeloid metaplasia with myelofibrosis (this includes all subtypes - chronic idiopathic myelofibrosis or angiogenic myeloid metaplasia, post thrombocythemic and post polycythemic myelofibrosis); patients must have anemia (hemoglobin < 11 g/dL) or palpable splenomegaly (measured in cm from costal margin - to be eligible); patients with palpable splenomegaly must have spleen size documented ultrasonographically as well; they must also meet standard diagnostic criteria for MMM
* Patients with morphologic evidence of advanced phases of the disease including accelerated (10-19% blasts) phase or with evidence of evolution to acute leukemia (>= 20% blasts) are also eligible for this study
* The Italian Diagnostic Criteria for MMM

  * Necessary criteria

    * Diffuse bone marrow fibrosis
    * Absence of the Philadelphia chromosome or BCR-ABL rearrangement in peripheral blood cells
  * Optional criteria

    * Splenomegaly of any grade
    * Anisopoikilocytosis with tear drop erythrocytes
    * Presence of circulating immature myeloid cells
    * Presence of circulating erythroblasts
    * Presence of clusters of megakaryoblasts and anomalous megakaryocytes in bone marrow sections
    * Myeloid metaplasia
  * Diagnosis of MMM is acceptable if the following combinations are present

    * The two necessary criteria plus any other two optional criteria when splenomegaly is present OR
    * The two necessary criteria plus any other four optional criteria when splenomegaly is absent
* Patients may have had prior chemotherapy or radiation therapy including splenic irradiation; prior therapy with erythropoietin, granulocyte-colony stimulating factor (GCSF), other growth factors or androgenic steroids is also permitted; there is no limit to the number of prior regimens received; at least 4 weeks must have elapsed since prior chemo or radiation therapy; at least 2 weeks must have elapsed since growth factor (erythropoietin, GCSF, granulocyte-macrophage colony-stimulating factor [GM-CSF]) or other therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 2mg/dL

  * In patients with associated hemolytic anemia; total bilirubin > 2mg/dL is permissible as long as this is as a result of predominantly unconjugated hyperbilirubinemia; such patients may be enrolled only after discussion with the study chair
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal unless due to disease
* Serum creatinine =< 2mg/dL
* Patients must not be pregnant or nursing; women of child- bearing potential and men must agree to use an effective contraceptive method; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior therapy with decitabine
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) disease should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with decitabine
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-09-29 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi M Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (14):
- United States (14):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lin C, Patel AA, Huo D, Karrison T, van Besien K, Godwin J, Sher D, Weiner H, Green M, Wade JL 3rd, Klisovic R, Baer MR, Larson RA, Stock W, Odenike O. A multicenter phase 2 clinical trial of low-dose subcutaneous decitabine in myelofibrosis. Blood Adv. 2024 Nov 26;8(22):5735-5743. doi: 10.1182/bloodadvances.2024013215. PMID 39250708

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine: Patients receive 0.3 mg/kg/day decitabine subcutaneously on days 1-5 and 8-12.
  decitabine : Given SC
Period: Overall Study
Arm/Group | Decitabine
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients receive 0.3 mg/kg/day decitabine subcutaneously on days 1-5 and 8-12.
  decitabine : Given SC
Arm/Group | Arm I
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response, Partial Response, or Hematologic Improvement.
Description: Complete response is normalization of counts and transfusion-independence.
  Partial response is hemoglobin increase to normal levels, multilineage improvement including absolute neutrophil count (ANC) and/or platelets.
  Hematologic improvement is red cell transfusion-independence or >50% increase in platelet levels.
Time Frame: Up to 36 weeks (6 cycles)
Population: Two patients were non-evaluable for response.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I
Number analyzed (Participants) | 19
percentage of participants | 37 [17 to 54]

2. Primary Outcome: Incidence of Toxicities, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0
Description: Percentage of patients experiencing any toxicity, any grade level. Additional details on adverse events are reported in Adverse Events section.
Time Frame: Up to 30 days of last dose of decitabine
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm I: Patients receive decitabine subcutaneously on days 1-5 and 8-12.
  decitabine: Given SC
Arm/Group | Arm I
Number analyzed (Participants) | 21
percentage of patients | 100 [84 to 100]

3. Secondary Outcome: CD34+ Cells
Description: CD34 positive(+) cells are determined by flow immunostaining and light scatter in peripheral blood. Samples are then analyzed by flow cytometry, and CD34+ cells quantitated after 75,000 CD45 events are studied. (At least 75,000 CD45 events must be studied to ensure accuracy of the assay). Absolute numbers are determined by multiplying the % CD34+ cells by the total white blood cell count obtained on a CBC that is processed simultaneously.
Time Frame: Cycle 1, Day 1
Population: One patient had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 20
cells x 10^6/L | 117 [44 to 310]

4. Secondary Outcome: CD34+ Cells
Description: as for outcome 3
Time Frame: Cycle 1, Day 5
Population: One patient had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 20
cells x 10^6/L | 71 [31 to 159]

5. Secondary Outcome: CD34+ Cells
Description: as for outcome 3
Time Frame: Cycle 1, Day 12
Population: Three patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 18
cells x 10^6/L | 35 [14 to 88]

6. Secondary Outcome: CD34+ Cells
Description: as for outcome 3
Time Frame: Cycle 2, Day 1
Population: Five patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 16
cells x 10^6/L | 76 [23 to 243]

7. Secondary Outcome: CD34+ Cells
Description: as for outcome 3
Time Frame: Cycle 2, Day 5
Population: Six patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 15
cells x 10^6/L | 35 [14 to 87]

8. Secondary Outcome: CD34+ Cells
Description: as for outcome 3
Time Frame: Cycle 2, Day 12
Population: Six patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: cells x 10^6/L
Arm/Group | Arm I
Number analyzed (Participants) | 15
cells x 10^6/L | 21 [8 to 58]
Statistical Analysis 1: Comparison: Arm I; Mixed effects regression analysis of change over time in CD34+ cell levels. Analysis performed on log scale; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; 5 degrees of freedom test over six time points: day 1 (pre-treatment) and days 5, 12, 43, 47, and 54 post treatment

9. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 1, Day 1
Population: Four patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 17
ratio | 4.4 [2.6 to 7.3]

10. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 1, Day 5
Population: Three patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 18
ratio | 5.7 [4.1 to 8.0]

11. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 1, Day 12
Population: Three patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 18
ratio | 6.4 [4.0 to 10.1]

12. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 2, Day 1
Population: Seven patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 14
ratio | 4.0 [2.4 to 6.8]

13. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 2, Day 5
Population: Seven patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 14
ratio | 6.0 [3.7 to 9.6]

14. Secondary Outcome: CXCR4
Description: CXCR4 gene expression level measured by real-time RT_PCR. Ratio of CXCR4 vs a housekeeping gene (i.e., ABL)
Time Frame: Cycle 2, Day 12
Population: Eleven patients had missing data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Arm I
Number analyzed (Participants) | 10
ratio | 7.1 [3.8 to 13.1]
Statistical Analysis 1: Comparison: Arm I; Mixed effects regression analysis of change over time in CXCR4 levels. Analysis performed on log scale; Test type: Superiority or Other; p = 0.29, Mixed Models Analysis; 5 degrees of freedom test over six time points: day 1 (pre-treatment) and days 5, 12, 43, 47, and 54 post treatment

15. Secondary Outcome: Hemoglobin F
Description: Percentage of hemoglobin F as a proportion of total Hb (%HbF) measured by HPLC on peripheral blood samples.
  Midpoint of 0.5% imputed for values reported as below limit of detection (1.0%). Hemoglobin F has been previously shown to be upregulated by decitabine in other hematologic disorders- sickle cell disease specifically. The rationale for exploring it in this study was to evaluate its potential utility as a biomarker of drug effect/PD marker.
Time Frame: Cycle 1, Day 1
Population: Four patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 17
percentage of HbF | 1.6 [0.8 to 2.5]

16. Secondary Outcome: Hemoglobin F
Description: as for outcome 15
Time Frame: Cycle 1, Day 5
Population: Three patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 18
percentage of HbF | 1.6 [0.7 to 2.5]

17. Secondary Outcome: Hemoglobin F
Description: as for outcome 15
Time Frame: Cycle 1, Day 12
Population: Three patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 18
percentage of HbF | 1.4 [0.6 to 2.2]

18. Secondary Outcome: Hemoglobin F
Description: as for outcome 15
Time Frame: Cycle 2, Day 1
Population: Nine patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 12
percentage of HbF | 1.5 [0.5 to 2.5]

19. Secondary Outcome: Hemoglobin F
Description: as for outcome 15
Time Frame: Cycle 2, Day 5
Population: Seven patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 14
percentage of HbF | 1.5 [0.6 to 2.4]

20. Secondary Outcome: Hemoglobin F
Description: as for outcome 15
Time Frame: Cycle 2, Day 12
Population: Seven patients had missing data.
Measure: Mean (95% Confidence Interval); unit: percentage of HbF
Arm/Group | Arm I
Number analyzed (Participants) | 14
percentage of HbF | 1.5 [0.8 to 2.2]
Statistical Analysis 1: Comparison: Arm I; Mixed effects regression analysis of change over time in hemoglobin F levels; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis; 5 degrees of freedom test over six time points: day 1 (pre-treatment) and days 5, 12, 43, 47, and 54 post treatment

ADVERSE EVENTS:
Time Frame: Up to 30 days of last dose of decitabine
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 15/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=21)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Blood (Infections and infestations) | 3
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Catheter-related (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Lung (pneumonia) (Infections and infestations) | 2
Splenic infarct vs hemorrhage/rupture (Vascular disorders) | 1
Sweet's Syndrome (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Confusion (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Fever (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 1
Hematoma (Vascular disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 4
Oesophageal varices (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 3
Urinary retention (Renal and urinary disorders) | 1
Vascular disorders - Other (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=21)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 8
Anemia (Blood and lymphatic system disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
CD4 lymphocytes decreased (Investigations) | 2
Chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine increased (Investigations) | 5
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Fever (General disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 4
INR increased (Investigations) | 4
Infections and infestations - Other (Infections and infestations) | 5
Injection site reaction (General disorders) | 2
Insomnia (Psychiatric disorders) | 2
Lymphocyte count decreased (Investigations) | 3
Mucositis oral (Gastrointestinal disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 7
Neutrophil count decreased (Investigations) | 15
Oral hemorrhage (Gastrointestinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Platelet count decreased (Investigations) | 16
Proteinuria (Renal and urinary disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Urinary frequency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less